CLINICAL TRIAL: NCT02259205
Title: Cardio Protective Properties of a Yogurt Enriched With Bioactive Lipids of Olive Oil Products
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harokopio University (Other)
Collaborators: National and Kapodistrian University of Athens (Other); Competitiveness and Entrepreneurship (OPCE II), NRSF 2007-13 (Unknown)
Responsible Party: Principal Investigator, Smaragdi Antonopoulou, Professor in Biochemistry, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 11SYN-2-652; HUA (Other: HUA)
Record Dates: First submitted 2014-09-24; First posted 2014-10-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Cardiovascular Diseases
Keywords: platelet activating factor; inflammatory markers; yogurt; olive oil; platelet aggregation; oxidative stress; endothelial damage; bioactive lipids
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Enriched Yogurt (Experimental): 150 g yogurt enriched with approximately 0.5 g bioactive lipids extract from olive oil mill provided daily for 8 weeks
  Interventions: Other: Enriched Yogurt
- Plain Yogurt (Placebo Comparator): 150 g not enriched yogurt provided daily for 8 weeks
  Interventions: Other: Plain Yogurt
- Control (No Intervention): No yogurt consumption

INTERVENTIONS:
Other: Enriched Yogurt — 150 g yogurt enriched with bioactive lipids extract from olive oil mill will be provided daily for 8 weeks
  Arms: Enriched Yogurt
Other: Plain Yogurt — 150 g plain yogurt will be provided daily for 8 weeks
  Arms: Plain Yogurt

SUMMARY:
This study evaluates the effectiveness of a yogurt enriched with bioactive lipids extracted from olive mill waste in platelet aggregation and other inflammatory and oxidative stress markers. The study will include three groups: the intervention group will receive the enriched yogurt while the other two groups will serve as controls (plain yogurt and no yogurt consumption).

DETAILED DESCRIPTION:
Cardiovascular diseases are the leading cause of mortality worldwide. Data from the investigators research group indicate that platelet activating factor (PAF) is one of the most important inflammatory factors and the main mediator of thrombosis during the formation of atherosclerotic plaque. Thus, dietary interventions aimed at inhibition of PAF is of particular importance in public health level. The aim of the study is to examine the efficacy of administering in humans bioactive lipids extracted from olive mill waste (with proven in vitro anti-thrombotic activity and in vivo anti-atherosclerotic properties in rabbits fed an atherogenic diet) to inhibit the activity of PAF and other inflammatory mediators.

Bioactive lipids are isolated by standardized methodology of oil manufacture byproducts. Preliminary studies have been done in animals to establish the safety of administration of these compounds and to clarify the effective dosages of administration for inhibiting formation of atherosclerotic plaques. The effectiveness of these compounds in humans will be examined in a randomized, double-blind clinical trial in subjects aged 40-60 years, lasting eight weeks. Supplementation with the bioactive lipids will be in the form of an enriched yogurt provided daily. The study includes three groups: treatment group, where enriched yogurt will be provided, plain yogurt treatment group and no consumption of yogurt group . Parameters that will be assessed are the inhibition of platelet aggregation (with three different stimuli, including PAF), lipid profile, inflammatory markers such as CRP, IL-6, TNFa, and oxidative stress markers.

ELIGIBILITY:
Inclusion Criteria:

* All individuals, aged 40-60 years, without any of the exclusion criteria

Exclusion Criteria:

* Any anti-inflammatory medication
* Hyper-lipidemic medications
* Use of antibiotics within two months from study entry
* Pregnancy or childbirth in the previous year
* Intake of any nutritional supplement
* Any serious dental, respiratory, liver, kidney, gastrointestinal disease

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-07 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Changes in Platelet aggregation | 0 (baseline), end of 4th week and 8th week
  The ability of platelets to aggregate will be measured in platelet rich plasma (PRP) of volunteers using PAF, thrombin and ADP as aggregating factor.

SECONDARY OUTCOMES:
Changes in Blood lipid profile | 0 (baseline), end of 4th week and 8th week
  Blood levels of cholesterol, LDL-cholesterol, HDL-cholesterol and triacylglycerols will be measured.
Changes in Glucose and Insulin | 0 (baseline), end of 4th week and 8th week
  Blood levels of glucose and insulin
Changes in Gastro-intestinal symptoms | 0 (baseline), end of 4th week and 8th week
  Gastro-intestinal symptoms and possible side effects from yogurt consumption will be assessed through validated questionnaires.
Change in Dietary intake | 0 (baseline), end of 8th week
  Dietary intake will be assessed through two dietary recalls and a food frequency questionnaire at each time point.
Changes in Oxidative stress | 0 (baseline), end of 4th week and 8th week
  Ex vivo serum oxidation as a marker for lipid oxidation and protein carbonyls as a marker for protein oxidation will be measured.
Changes in Gut microbiota populations | 0 (baseline), end of 8th week
  the populations of lactobacilli, bifidobacteria and Clostridium histolyticum group will be estimated by real-time PCR using genus specific primers. Furthermore, the metabolic products of the gut microorganisms will be evaluated by measuring the short chain fatty acids profile in fecal samples.
Changes in Inflammation-related markers | 0 (baseline), end of 4th week and 8th week
  C-reactive protein (CRP), IL-6, TNFa, IL-10 levels in fasting blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Smaragdi Antonopoulou, PhD, Principal Investigator — Harokopio University, Department of Nutrition and Dietetics; Elizabeth Frafopoulou, PhD, Study Chair — Harokopio University, Department of Nutrition and Dietetics; Tzortzis Nomikos, PhD, Study Chair — Harokopio University, Department of Nutrition and Dietetics
Locations (1):
- Harokopio University, Department of Nutrition and Dietetics, Athens, Attica, Greece

REFERENCES:
- [Derived] Antonopoulou S, Mitsou EK, Kyriacou A, Fragopoulou E, Detopoulou M. Does Yogurt Enriched with Platelet-Activating Factor Inhibitors from Olive Oil By-Products Affect Gut Microbiota and Faecal Metabolites in Healthy Overweight Subjects? (A randomized, parallel, three arm trial.). Front Biosci (Landmark Ed). 2024 Apr 23;29(4):159. doi: 10.31083/j.fbl2904159. PMID 38682205
- [Derived] Detopoulou M, Ntzouvani A, Petsini F, Gavriil L, Fragopoulou E, Antonopoulou S. Consumption of Enriched Yogurt with PAF Inhibitors from Olive Pomace Affects the Major Enzymes of PAF Metabolism: A Randomized, Double Blind, Three Arm Trial. Biomolecules. 2021 May 28;11(6):801. doi: 10.3390/biom11060801. PMID 34071485